CLINICAL TRIAL: NCT05513898
Title: Treatment of Pilonidal Cyst With Holmium Laser
Acronym: PILOLAS
Status: Completed | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: COS-RGDS-2020-06-028-
Record Dates: First submitted 2022-06-23; First posted 2022-08-24 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Pilonidal Cyst
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational study on the treatment of pilonidal cyst with Holmium laser. Single-centre retrospective study of medical data from patients' medical records

DETAILED DESCRIPTION:
From the medical records of a series of patients treated for pilonidal cysts with Holmium laser:

1. Primary objective: to assess the rate of healing at 1 month after Holmium laser treatment (healing being defined as no dressing)
2. Secondary objectives: to assess the following:

   * Healing rate at last follow-up (1 month after surgery)
   * Recurrence rate at last follow-up (1 month after surgery)
   * Consumption of >1 level analgesics in the week and month following the procedure
   * Duration of nursing care

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older, who has been informed of the research;
* Patient with a pilonidal cyst treated with Holmium Laser during a scheduled procedure.

Exclusion Criteria:

* Patient under legal protection, guardianship or curatorship;
* Patient who has indicated his opposition to the use of his data.
* Patient undergoing emergency surgery for an abscess

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients participating in the study were operated on at the centre between AUGUST and NOVEMBER 2020. The study is based solely on a review of the medical records of these patients. No further evaluation is planned.
Sampling Method: Non-Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Healing rate | Month 1
  explanatory analysis of the healing rate at Month 1

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique de la Sauvegarde, Lyon, France

IPD SHARING:
Plan to Share IPD: No